CLINICAL TRIAL: NCT05273671
Title: Comparison Between Nalbuphine Versus Dexmedetomidine for Prevention of Emergence Agitation in Pediatrics During Sevoflurane Anesthesia: Prospective Randomized Controlled Clinical Trial
Brief Title: Nalbuphine Versus Dexmedetomidine for Prevention of Emergence Agitation in Pediatrics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0305447
Record Dates: First submitted 2022-02-19; First posted 2022-03-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Nalbuphine; Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: allocated children will be randomly assigned through computer-generated random numbers contained in sealed opaque envelopes to one of the three groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nalbuphine (Experimental): 0.1 mg/kg nalbuphine diluted in 10 ml I.V 10 minutes before the end of surgery
  Interventions: Drug: Nalbuphine
- dexmedetomedine (Experimental): receive dexmedetomedine 0.5 mic/kg diluted in 10 ml I.V 10 minutes before the end of surgery
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator): receive a saline solution 10 min before the end of surgery
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Nalbuphine — will receive 0.1 mg/kg NAL diluted in 10 ml I.V 10 minutes before the end of surgery
  Other Names: nalophen
  Arms: nalbuphine
Drug: Dexmedetomidine — will receive dexmedetomedine 0.5 mic/kg diluted in 10 ml I.V 10 minutes before the end of surgery
  Other Names: Precedex
  Arms: dexmedetomedine
Drug: normal Saline — will receive with a saline solution 10 min before the end of surgery
  Other Names: saline
  Arms: saline

SUMMARY:
the investigators hypothesized that Nalbuphine may be alternative pharmacological agent for prevention of emergence agitation in pediatrics who will be scheduled for elective lower abdominal surgical procedures (inguinal hernia repair and hypospadias) during sevoflurane anesthesia

DETAILED DESCRIPTION:
SEVOFLURANE is widely used popular inhalational anesthetic to induce and maintain anesthesia in children due to its greater hemodynamic stability, less irritation of the airway and low blood gas solubility coefficient, which causes rapid emergence and recovery from general anesthesia in pediatric anesthesia. [1] However, sevoflurane anesthesia is frequently associated with emergence agitation (EA) in children with incidence ranging up to 80%. [2-5] EA is a complex phenomenon and a variety of explanations have been proposed for its etiology. These include multiple surgical and patient related factors as well as anesthesia related factors such as rapid emergence due to the low blood solubility of sevoflurane.[1,2,6] Despite it is usually self limited; EA is still a considerable side-effect because of the risks of falling, self-injury to the child or to the surgical site, the stress caused to both caregivers and families, moreover, increase the need for continuous monitoring of patients by recovery room staffs and physical restraint of patient.[6] Several medications like propofol, fentanyl, a2-adrenergic receptor agonist and ketamine have been investigated in an attempt to reduce the occurrence and severity of EA, with variable outcomes. [4-11] Dexmedetomidine is an a-2 adrenergic agonist with a larger ratio of a2/a1 activity (1600:1) when compared to clonidine (200:1).The hemodynamic effects of dexmedetomidine are similar to that of clonidine and the effects can vary depending on the dose, rat. [10] Nalbuphine (NAL) is a synthetic opioid agonist antagonist acts on kappa and mu opioid receptor producing analgesia and sedation .One of the advantages of NAL over pure narcotic agonists is inducing minimal respiratory depression, it is considered a safe drug and the large margin of safety make it often used for pediatric patients. It has been shown that the use of nalbuphine carries a lower risk of adverse events like nausea, vomiting, pruritus, constipation, and respiratory depression Our primary outcome: The incidence of post-operative EA Secondary outcome:Time to emergence in minutes Time to extubation in minutes Children's hospital eastern Ontario pain scale. Discharge time (min) The time of first postoperative analgesic dose Possible postoperative side effects. All patients will undergo thorough preoperative evaluation, which include history, physical examination and relevant laboratory investigations. None of the patients will be given any solid food for 6 hours preoperatively but each will be encouraged to take clear fluids until 2 hours before induction of anesthesia. All patients will be pre-medicated with 0.3 mg/kg oral midazolam (maximum dose of 12 mg) 30 min before induction. Upon arrival at the operating room, patients will be monitored by non-invasive the blood pressure, temperature, electrocardiogram capnography and pulse oximetry.

Inhalation induction will be done via transparent face mask after saturating the breathing system (Jackson-Rees modification of Ayer's T-piece) with a mixture of sevoflurane 8 vol % in 100% O2 (6 L/min). After loss of consciousness, intravenous line will be inserted and Rocuronium 0.6 mg/kg is administered and when adequate depth of anesthesia is reached, a laryngeal mask airway (LMA) of appropriate size for the age and weight of the child will be placed .Anesthesia will maintained with sevoflurane at 2 3 vol % in 40% O2 in air to maintain a stable heart rate, blood pressure and respiratory rate (base line ± 20%). Paracetamol 15 mg/kg (Perfalgan® 100 ml vial UPSA France) and Dexamethasone 0.3 mg/kg will be administered IV to each child immediately after the induction of anesthesia. Lung ventilation will be controlled to maintain the end tidal carbon dioxide tension between 30 and 35 mmHg. Caudal block with 1.0 ml/kg 0.25% bupivacaine will be performed in all patients. Failure of caudal block will be defined as increase in heart rate and or mean arterial blood pressure (MAP) > 10% than pre-incisional value at the start of surgery. No opioid will be given; no propofol will be used during the procedure.

The allocated children will be randomly assigned through computer-generated random numbers contained in sealed opaque envelopes to one of the three groups:

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I &II
* scheduled for elective lower abdominal surgical procedures (inguinal hernia repair and hypospadias) under general anesthesia

Exclusion Criteria:

* history of hypersensitivity to the studied drug,
* refusal of the legal guardian
* chronic or acute intake of any sedative or analgesic drugs,
* Psychological& emotional disorder.
* Cognitive or developmental disorders.
* severely agitated child at induction of anesthesia
* Any neurological condition that would limit the patient's ability to communicate with or understand nursing personnel,
* Existing contraindications to caudal block such as coagulopathy, local and systemic infection.
* Failure of the caudal block.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-02 (Estimated)

PRIMARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) change | at 5, 10, 20 and 30 minutes post-operatively
  Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) based on crying, facial expression, verbal statements, position of torso, touching of the wound and movement of legs will be used for post-operative pain assessment
  * minimum score: 4 best
  * maximum score: 13 worse
pediatric anesthesia emergence delirium (PAED) scale change | at 5, 10, 20 and 30 minutes post-operatively
  pediatric anesthesia emergence delirium (PAED) scale, scale that define the child's behavior in the recovery room
  1. sleeping (best)
  2. awake, calm
  3. irritable, crying
  4. inconsolable crying (worse)

SECONDARY OUTCOMES:
The time of first postoperative analgesic dose | up to 24 hours post operative
  in minutes

OTHER OUTCOMES:
occurrence of side effects in PACU like nausea and vomiting. | up to 24 hours post operative
  incidence and severity

CONTACTS AND LOCATIONS:
Overall Officials: yasser M osman, Principal Investigator — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No